CLINICAL TRIAL: NCT00833365
Title: Early vs. Late Use of Ibuprofen for Patent Ductus Arteriosus (PDA) Closure and Pain/Stress Reduction
Brief Title: Early Versus Late Use of Ibuprofen for Patent Ductus Arteriosus (PDA) Closure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study drug not available
Sponsor: University of Utah (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31394
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Results first posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2014-12

CONDITIONS: Patent Ductus Arteriosus; Prematurity
Keywords: premature infants; PDA; ibuprofen
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early treatment (Active Comparator): Infants randomized to this group will receive their initial dose of ibuprofen prior to reaching 96 hrs old
  Interventions: Drug: Ibuprofen
- Late treatment (Active Comparator): Infants randomized to this group will receive their initial dose of ibuprofen after infant has reached 96 hrs old but before the infant reaches 10 days old.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen 10 mg/kg/dose for one dose, then repeated 24 hrs later at 5 mg/kg/dose and repeated 24 hrs later at 5 mg/kg/dose
  Other Names: NeoProfen
  Arms: Early treatment
Drug: Ibuprofen — Initial dose of ibuprofen is 10 mg/kg and then repeated every 24 hours times two with doses of 5 mg/kg
  Other Names: NeoProfen
  Arms: Late treatment

SUMMARY:
The primary objective is to evaluate the Patent Ductus Arteriosus (PDA) closure rate of early vs. late use of Ibuprofen (Ibu). The investigators believe that early use of Ibu will have a higher PDA closure rate than later use of Ibu. Early use is defined as medication given before the infant reaches 96 hrs old. Late use is defined as medication given when infant is more than 96 hrs old.

DETAILED DESCRIPTION:
Infants with birth weight at <1200gm and/or <28 weeks gestation who have been diagnosed with a Patent Ductus Arteriosus (PDA) qualify for the study if there are no contraindications to treatment. Infants are randomized into treatment arms of <96 hrs old and >96 hrs old. Ibuprofen is given in the dosage of 10 mg/kg on initial dose, followed 24 hours later by 5 mg/kg dose and then 24 hours later another dose of 5 mg/kg. An echocardiogram will be done prior to treatment and then within 48 hours after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight less than 1200gm
* Less than 28 weeks gestational age
* Confirmed Patent Ductus Arteriosus (PDA) via echocardiogram and clinical exam

Exclusion Criteria:

* Active Bleeding
* Currently being treated for Persistent Pulmonary Hypertension (PPHN)
* Cardiac anomalies
* Chromosomal abnormalities
* Endocrine, metabolic, renal, or hepatic disorders

Max Age: 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Chan, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Treatment | Late Treatment
Started | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Treatment | Late Treatment | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 6 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of PDA Closures Related to Treatment With Ibuprofen
Description: Closure of the Patent Ductus in response to early or late treatment of ibuprofen was evaluated by echocardiogram. There is only one event (closure) possible per participant.
Time Frame: Within 48 hrs of ibuprofen round
Population: Premature infants born at 23+3 weeks to 29+4 weeks with positive patent ductus arteriosus on cardiac echogram were randomized to early or late treatment with ibuprofen. 2 babies which had been originally randomized to the late treatment arm never got ibuprofen and are not included in analysis.
Measure: Number; unit: closures related to treatment
Arm/Group | Early Treatment | Late Treatment
Number analyzed (Participants) | 9 | 4
closures related to treatment | 1 | 0

2. Secondary Outcome: Plasma Catecholamines, Glucose, and Lactate Levels 1 and 6 Hours After Ibuprofen Administration
Time Frame: 1 and 6 hours
Population: Due to early termination of the study, labs were not analyzed.
Arm/Group | Early Treatment | Late Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Early Treatment | Late Treatment
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Treatment (N=9) | Late Treatment (N=6)
Death (Infections and infestations) | 1 | 0 — Infant died from necrotizing enterocolitis, an abdominal infection not unexpected in the premature infant population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No